CLINICAL TRIAL: NCT01201239
Title: An Open Pilot Study to Evaluate the Efficacy and Safety, Tolerability of Raltegravir（RAL）in Treatment-experienced HIV-1 Infected Adult Chinese Patients
Brief Title: Efficacy and Safety of Raltegravir (RAL) in Treatment-experienced HIV-1 Infected Adult Chinese Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Hongzhou Lu, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAL-001
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: HIV
Keywords: raltegravir; HIV-1; drug resistance
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- raltegravir (Experimental): HIV-infected patients aged over 18 who have failed previous antiretroviral treatment with multi-drug resistant or with multi-drug intolerance are to accept Ral plus OBT.
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — RAL 400 mg twice daily plus OBT (optimized background therapy) for 48 weeks

SUMMARY:
To assess the safety, tolerability and efficacy of Raltegravir (RAL) when combined with other antiretroviral drugs in treatment-experienced Chinese HIV-infected patients, including those with multi-drug resistant HIV-1 infection or drug intolerance.

DETAILED DESCRIPTION:
An open, prospective, uncontrolled pilot study to evaluate the efficacy and safety of raltegravir in treatment-experienced HIV-1 infected adult patients who have failed the previous antiretroviral treatment due to drug resistance or drug intolerance.

1. Patients Enrollment:

   HIV-infected patients aged over 18 who have failed previous antiretroviral treatment with multi-drug resistant or with multi-drug intolerance are eligible. And at least 50 subjects are to be concluded in the trial.

   ⅰ) The diagnostic criteria of HIV/AIDS refer to guidelines for diagnosis and treatment of HIV/AIDS in China(2005).

   ⅱ) Treatment failure will be defined as follows: (i): HIV viral load has decreased by less than 1 log copies/ml in patients with 8 weeks of HAART, or (ii) HIV viral load is still detectable after 6 months of HAART;or (iii) reappearance of a detectable viral load after HAART has led to undetectable viral load.

   ⅲ) The definition of drug resistance is based on a genotypic resistance test.

   ⅳ) Drug intolerance involves all the serious antiretroviral drug related adverse events, such as AZT related bone marrow suppression, NVP or EFV related serious liver damage and allergic reaction, d4T related lactic acidosis, pancreatitis and peripheral neuritis, etc.
2. Patients enrolled in the study sign consent form.
3. Antiretroviral regimen for the subjects:

   The patients enrolled in the study accept a treatment regimen of RAL 400 mg twice daily plus OBT (optimized background therapy), which is selected on the basis of the patient's antiretroviral treatment history, results from all available genotypic resistance tests, previous or current laboratory abnormalities and intolerance to other antiretroviral drugs, and shall, if possible, contain two anti-retroviral drugs fully active against the patient's virus by genotype.
4. Data collection:

   For each patient, detection of HIV viral load and CD4+ T lymphocyte count is done at screening, and at weeks 4, 12, 24 and 48. The safety profile of RAL is monitored according to patients' complaints and the results of physical and laboratory examinations. Plasma HIV RNA viral loads are determined by HIV-1 Quantiplex(bDNA) assay approved by FDA. CD4+ T lymphocytes are counted with flow cytometry. Any drug-related adverse events that patients experience during treatment will be recorded, such as nausea, vomiting, abdominal pain, abodominal distension, diarrhea, fever, headache, dizzy, fatigue etc. Laboratory examinations cover blood, urine and stool routine, liver and renal function, electrolytes, blood glucose, blood lipid, electrocardiogram etc.
5. Endpoints of study:

The primary endpoint is the the safety and tolerability of RAL 400 mg b.i.d. in combination with OBT, assessed by review of the accumulated safety data in HIV-infected adult patients. The secondary endpoint is antiretroviral activity of RAL 400 mg b.i.d. in combination with OBT as measured by change at week 24 in viral load from baseline, increase of CD4+ T lymphocytes compared to baseline and proportions of patients with: viral load less than 400 copies/ml; viral load less than 50 copies/ml; and a reduction in viral load from baseline exceeding 1.0 log10 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients aged over 18 who have failed previous antiretroviral treatment with multi-drug resistant or with multi-drug intolerance

Exclusion Criteria:

* The patient is aged below 18 or over 65 years
* The patient has serious opportunistic infections or tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
the safety and tolerability of RAL 400 mg b.i.d. in combination with optimized background therapy (OBT), assessed by review of the accumulated safety data in HIV-infected adult patients. | 48 weeks

SECONDARY OUTCOMES:
antiretroviral activity of RAL 400 mg b.i.d. in combination with OBT as measured by change at week 24 in viral load from baseline, increase of CD4+ T lymphocytes compared to baseline | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China